CLINICAL TRIAL: NCT05392114
Title: An Open-Label, Long Term Safety and Efficacy Study of Donidalorsen in the Prophylactic Treatment of Hereditary Angioedema (HAE)
Brief Title: A Study to Assess the Long-Term Safety and Efficacy of Donidalorsen in the Prophylactic Treatment of Hereditary Angioedema (HAE)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 721744-CS7; 2022-000757-93 (EudraCT Number)
Expanded Access: NCT06415448 (Available)
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedema
Keywords: HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — donidalorsen; IONIS-PKK-LRx

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OLE Participants (Experimental): Group 1 and Group 2 participants will be administered donidalorsen by SC injection for up to 157 weeks.
  Interventions: Drug: Donidalorsen

INTERVENTIONS:
Drug: Donidalorsen — Donidalorsen will be administered by SC injection.
  Other Names: ISIS 721744; IONIS-PKK-LRx

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of donidalorsen in people with HAE and the effects of donidalorsen on the number of HAE attacks and their impact on quality of life (QoL).

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, open-label, global study with donidalorsen in up to approximately 144 participants with HAE-1 (Type I) and HAE-2 (Type II). There are two groups in this study: 1) participants who roll over from another study of donidalorsen (open-label extension [OLE] participants), and 2) new participants who are not rolling over from another study of donidalorsen and were previously maintained on HAE prophylactic therapy with lanadelumab, berotralstat, or a C1-esterase inhibitor (C1-INH). The length of participation in the study is approximately 70 weeks for OLE participants and 76 weeks for other participants. Participants will receive donidalorsen in an Extended Treatment Period for up to an additional 104 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Participants and, as applicable, legally authorized representatives (i.e., parent(s)/legal guardian), must provide written and signed informed consent form (ICF).
2. Participants must have access to, and the ability to use, ≥ 1 acute medication(s) (e.g., plasma-derived or recombinant C1-INH concentrate or a bradykinin receptor (BK) 2-receptor antagonist) to treat angioedema attacks.

   Open-Label Extension Participants ONLY:
3. Satisfactory completion of ISIS 721744-CS5 (randomized placebo-controlled index study) through Week 25 or participants who are allowed to exit ISIS 721744-CS5 study per protocol with an acceptable safety and tolerability profile.

   New (not previously on donidalorsen) Participants ONLY:
4. Participants must be aged ≥ 12 years at the time of informed consent and, as applicable, assent.
5. Participants must have a documented diagnosis of HAE-1/HAE-2.
6. Participants must be on a stable dose (≥ 12 weeks) of prophylaxis treatment with lanadelumab or berotralstat or SC C1-esterase inhibitor prior to the Screening Period.

Exclusion Criteria

Open-Label Extension Participants:

1. Have any new condition or worsening of an existing condition or change or anticipated change in medication.

   New (not previously on donidalorsen) Participants ONLY:
2. Concurrent diagnosis of any other type of recurrent angioedema, including acquired, idiopathic angioedema or HAE with normal C1-INH (also known as HAE Type III).
3. Anticipated change in the use of concurrent androgen or tranexamic acid prophylaxis used to prevent angioedema attacks.
4. Any clinically-significant abnormalities in screening laboratory values.
5. Malignancy within 5 years of Screening, except for non-melanoma skin cancers, cervical in situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma that has been successfully treated.
6. Hypersensitivity to the active substance (donidalorsen) or to any of the excipients.
7. Treatment with another investigational drug (non-oligonucleotide) or biological agent within 1 month of Screening or 5 half-lives of investigational agent, whichever is longer.
8. Recent history of, or current drug or alcohol abuse.
9. Participated in a prior donidalorsen study.
10. Exposure to any of the following medications:

    1. Angiotensin-converting enzyme (ACE) inhibitors or any estrogen containing medications with systemic absorption.
    2. Oligonucleotides (including small interfering ribonucleic acid [siRNA]) within 4 months of Screening if single dose received, or within 12 months of Screening if multiple doses received. This exclusion does not apply to vaccines.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with at Least One Treatment-emergent Adverse Event (TEAE), Graded by Severity | Up to approximately 70 weeks, plus 104 weeks for Group 1; up to approximately 76 weeks, plus 104 weeks for Group 2

SECONDARY OUTCOMES:
Time-normalized Number of Investigator-confirmed HAE Attacks (per Month) | Week 1 to Week 157 for Group 1 and Group 2
Percentage of Investigator-confirmed HAE Attack-free Participants | Week 1 to Week 157 for Group 1 and Group 2
Time-normalized Number of Moderate or Severe Investigator-confirmed HAE Attacks (per Month) | Week 1 to Week 157 for Group 1 and Group 2
Number of Investigator-confirmed HAE Attacks Requiring Acute Therapy | Week 1 to Week 157 for Group 1 and Group 2
Angioedema Quality of Life (AE-QoL) Questionnaire Total Score | Up to 157 weeks for Group 1 and Group 2
  The AE-QoL questionnaire is a validated tool to assess symptom-specific health-related QOL impairment in participants suffering from recurrent angioedema. The AE-QoL is a self-administered questionnaire comprising 17 questions across 4 domains: functioning, fatigue/mood, fears/shame, and food. The responses are scored from 1 to 5 where, 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = very often. Total and domain scores range from 0 to 100, with higher scores indicating greater impairment.

CONTACTS AND LOCATIONS:
Locations (48):
- United States (16):
  - Ionis Investigative Site, Paradise Valley, Arizona
  - Ionis Investigative Site, La Jolla, California
  - Ionis Investigative Site, Santa Monica, California
  - Ionis Investigative Site, Walnut Creek, California
  - Ionis Investigative Site, Tampa, Florida
  - Ionis Investigative Site, Kansas City, Kansas
  - Ionis Investigative Site, Boston, Massachusetts
  - Ionis Investigative Site, Ann Arbor, Michigan
  - Ionis Investigative Site, Detroit, Michigan
  - Ionis Investigative Site, St Louis, Missouri
  - Ionis Investigative Site, Mooresville, North Carolina
  - Ionis Investigative Site, Cincinnati, Ohio
  - Ionis Investigative Site, Columbus, Ohio
  - Ionis Investigative Site, Hershey, Pennsylvania
  - Ionis Investigative Site, Dallas, Texas
  - Ionis Investigative Site, Murray, Utah
- Ionis Investigative Site, Edegem, Belgium
- Ionis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Ionis Investigative Site, Ottawa, Ontario
  - Ionis Investigative Site, Edmonton
- France (3):
  - Ionis Investigative Site, La Tronche
  - Ionis Investigative Site, Marseille
  - Ionis Investigative Site, Paris
- Germany (3):
  - Ionis Investigative Site, Berlin
  - Ionis Investigative Site, Frankfurt
  - Ionis Investigative Site, München
- Israel (3):
  - Ionis Investigative Site, Ashkelon
  - Ionis Investigative Site, Haifa
  - Ionis Investigative Site, Tel Aviv
- Italy (5):
  - Ionis Investigative Site, Catania
  - Ionis Investigative Site, Napoli
  - Ionis Investigative Site, Padua
  - Ionis Investigative Site, Palermo
  - Ionis Investigative Site, San Donato Milanese
- Netherlands (2):
  - Ionis Investigative Site, Amsterdam
  - Ionis Investigative Site, Groningen
- Ionis Investigative Site, Krakow, Poland
- Ionis Investigative Site, San Juan, Puerto Rico
- Spain (4):
  - Ionis Investigative Site, Barcelona
  - Ionis Investigative Site, Madrid
  - Ionis Investigative Site, Seville
  - Ionis Investigative Site, Valencia
- Turkey (Türkiye) (3):
  - Ionis Investigative Site, Altındağ
  - Ionis Investigative Site, Bornova
  - Ionis Investigative Site, Istanbul
- United Kingdom (3):
  - Ionis Investigative Site, Birmingham
  - Ionis Investigative Site, Bristol
  - Ionis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.

REFERENCES:
- [Derived] Riedl MA, Bernstein JA, Jacobs JS, Craig T, Banerji A, Perego F, Lumry WR, Wedner HJ, Gierer S, Manning ME, Bordone L, Treadwell S, Lin T, Newman KB, Yarlas A, Cohn DM. Donidalorsen Treatment of Hereditary Angioedema in Patients Previously on Long-Term Prophylaxis. J Allergy Clin Immunol Pract. 2025 Sep;13(9):2381-2389.e3. doi: 10.1016/j.jaip.2025.06.018. Epub 2025 Jul 17. PMID 40673861